CLINICAL TRIAL: NCT06444295
Title: Project THRIVE: Testing an App-based Early Intervention to Reduce Alcohol Use and PTSD After Sexual Assault
Brief Title: Testing the Impact of Thrive App Versions on Alcohol Use and Posttraumatic Stress After Recent Sexual Assault
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Emily Dworkin, Associate Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00016193; R01AA030541 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Stress Symptom; Alcohol Drinking; Alcohol Problem
Keywords: Sexual assault; Mobile health intervention
MeSH Terms: conditions — Alcohol Drinking; Alcohol-Related Disorders | interventions — Cognitive Restructuring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- No experimental components (Active Comparator): Participants are invited to use a version of the app for 21 days. Participants receive only the non-core intervention components and do not attend coaching calls.
  Interventions: Behavioral: Non-core intervention components
- Activities + Thoughts (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Activities and Thoughts app modules, but do not attend coaching calls.
  Interventions: Behavioral: Activity scheduling; Behavioral: Cognitive restructuring; Behavioral: Non-core intervention components
- Activities only (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Activities app module, but do not attend coaching calls.
  Interventions: Behavioral: Activity scheduling; Behavioral: Non-core intervention components
- Thoughts only (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Thoughts app module, but do not attend coaching calls.
  Interventions: Behavioral: Cognitive restructuring; Behavioral: Non-core intervention components
- Activities, Thoughts, & Coaching (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Activities and Thoughts app modules and attend coaching calls.
  Interventions: Behavioral: Activity scheduling; Behavioral: Cognitive restructuring; Behavioral: Coaching calls; Behavioral: Non-core intervention components
- Activities + Coaching (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Activities app module and attend coaching calls.
  Interventions: Behavioral: Activity scheduling; Behavioral: Coaching calls; Behavioral: Non-core intervention components
- Thoughts + Coaching (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the Thoughts app module and attend coaching calls.
  Interventions: Behavioral: Cognitive restructuring; Behavioral: Coaching calls; Behavioral: Non-core intervention components
- Coaching only (Experimental): Participants are invited to use a version of the app for 21 days. Participants receive the non-core intervention components in the app and attend coaching calls.
  Interventions: Behavioral: Coaching calls; Behavioral: Non-core intervention components

INTERVENTIONS:
Behavioral: Activity scheduling — Participants will engage in activity scheduling in the app (i.e., "Activities" module). On the first day of using the app, users will create a list of valued/important and avoided activities (e.g., spending time with friends, going to the gym), and then have the option to add alcohol protective behavioral strategies (e.g., adding ice to drinks, alternating alcoholic and nonalcoholic beverages) to activities that the user identifies as being likely to involve drinking. On subsequent days, users will be encouraged to complete at least one activity from their list.
  Arms: Activities + Coaching; Activities + Thoughts; Activities only; Activities, Thoughts, & Coaching
Behavioral: Cognitive restructuring — Participants will engage in cognitive restructuring in the app (i.e., "Thoughts" activities). Users first go through an activity involving the identification of maladaptive cognitions and create a list of their maladaptive cognitions. On subsequent days, they engage in a guided in-app activity involving cognitive restructuring of maladaptive cognitions from their list.
  Arms: Activities + Thoughts; Activities, Thoughts, & Coaching; Thoughts + Coaching; Thoughts only
Behavioral: Coaching calls — Participants will receive 10-20 minute weekly coaching calls during the app use period (4 total, including coaching provided in the enrollment call). All coaching calls will, at minimum, include a check-in, troubleshooting of technical issues, check-in about experience with symptom self-monitoring, and offers of referrals. Coaching calls in conditions involving activity scheduling will involve assistance with the Activities module. Coaching calls in conditions involving cognitive restructuring will involve assistance with the Thoughts module.
  Arms: Activities + Coaching; Activities, Thoughts, & Coaching; Coaching only; Thoughts + Coaching
Behavioral: Non-core intervention components — All participants, regardless of condition, will receive the following non-core THRIVE components.
  * 21 days of brief self-report surveys in the app assessing their PTSD symptoms and alcohol use in the prior 24 hours.
  * A banner in their app displaying rotating non-personalized encouraging messages from other users. All app users will have the option of submitting encouraging statements to be displayed to all other users. Statements will be vetted by study staff before posting.
  * Lists of referral options specific to each recruitment site via the "Resources" section of the app.
  * Answers to frequently asked questions about the study, the study consent form, and contact information for the study team via the "Information" section of the app.
  * One call with a study "point person" within the first week following randomization to ensure they were able to access the app and troubleshoot access issues

SUMMARY:
The goal of this study is to find the most effective and efficient version of the THRIVE app. The THRIVE app is the first app-based preventative intervention that has been found to reduce alcohol misuse and posttraumatic stress in people who have recently experienced sexual assault. In this trial, participants are randomly assigned to receive different versions of the THRIVE app to compare their impact. The THRIVE app is currently only available to participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have reached the legal age of majority in their current state of residence
* Be able to read and speak English fluently
* Own a smartphone that cannot be accessed by others while the study app is installed, or they agree to take steps to reduce the risk that someone else will access the study app
* Be an enrolled undergraduate or graduate student at a recruitment site at the time of screening, or if they are on summer break, plan to be enrolled in the upcoming fall term
* Reside in the same state as the recruitment site for most of the year
* Have experienced a sexual assault (i.e., unwanted and non-consensual attempted/completed sexual contact) within the past 12 weeks at the time of screening
* Report ≥1 past-month heavy drinking episode (i.e., 5+ drinks on a given day or 15+ drinks in a given week for participants assigned male at birth and 4+ drinks on a given day or 8+ drinks in a given week for participants assigned female or intersex at birth) at the time of screening
* Endorse elevated posttraumatic stress symptoms at screening (defined as a score above a pre-established cut point on a screening measure of PTSD).

Exclusion Criteria:

* Active psychosis
* Location outside of the US at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Past-month alcohol problems | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed using the 16-item Short Form Rutgers Alcohol Problem Index (S-RAPI). Minimum score = 0, maximum score = 64, higher scores mean greater severity of problems.
Past-month number of drinks | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed via the online Timeline Followback (TLFB)
Past-month number of drinking days | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed via the online Timeline Followback (TLFB)
Past-month peak drinks | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed via the online Timeline Followback (TLFB)
Past-month frequency of heavy episodic drinking | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed via the online Timeline Followback (TLFB)
Past-month posttraumatic stress symptom severity | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed using the PTSD Checklist (PCL-5) in relation to the index assault. Minimum score = 0, maximum score = 80, higher scores mean greater severity of posttraumatic stress.
Past-month provisional diagnosis of posttraumatic stress disorder | Baseline, 1 month, 3 months, 6 months, 9 months, 1 year
  Assessed using the PTSD Checklist (PCL-5) in relation to the index assault. Provisional posttraumatic stress disorder diagnosis is defined as a score greater than or equal to 31.

SECONDARY OUTCOMES:
Drug use & problems | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 (not including alcohol questions)
Cannabis use & problems | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Cannabis Use Disorder Identification Test - Revised (CUDIT-R). Minimum score = 0, maximum score = 32, higher scores indicate hazardous cannabis use/possible cannabis use disorder.
Depression | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Center for Epidemiologic Studies Depression Scale - 10 item version. Minimum score = 0, maximum score = 30, higher scores mean greater depressive mood symptoms
Anxiety | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Generalized Anxiety Disorder-7 scale. Minimum score = 0, maximum score = 21, higher scores indicate greater severity of generalized anxiety symptoms.

OTHER OUTCOMES:
Positive mental health | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Flourishing Scale. Minimum score = 8, maximum score = 56, higher scores indicate people with many psychological resources and strengths.
Flourishing | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Flourishing Index. Minimum score = 0, maximum score = 120, higher scores indicate greater levels of flourishing/human well-being in individuals.
Social support | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the Multidimensional Scale of Perceived Social Support. Minimum score = 12, maximum score = 84, higher scores indicate greater level of perceived social support.
Loneliness | Baseline, 3 months, 6 months, 9 months, 1 year
  Assessed using the University of California Los Angeles 3-Item Loneliness Scale. Minimum score = 3, maximum score = 9, higher scores indicate greater levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dworkin, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No